CLINICAL TRIAL: NCT05268016
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2a Study to Assess the Efficacy and Safety of ME3183 Administered Orally in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy and Safety of ME3183 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meiji Pharma USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ME3183-3
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ME3183 Dose 1, BID (Experimental): Specified dose of ME3183 capsule for 16 weeks
  Interventions: Drug: ME3183
- ME3183 Dose 2, QD (Experimental): Specified dose of ME3183 capsule for 16 weeks
  Interventions: Drug: ME3183
- ME3183 Dose 3, BID (Experimental): Specified dose of ME3183 capsule for 16 weeks
  Interventions: Drug: ME3183
- ME3183 Dose 4, QD (Experimental): Specified dose of ME3183 capsule for 16 weeks
  Interventions: Drug: ME3183
- Placebo (Placebo Comparator): Placebo capsule of ME3183 for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ME3183 — ME3183 capsule
  Arms: ME3183 Dose 1, BID; ME3183 Dose 2, QD; ME3183 Dose 3, BID; ME3183 Dose 4, QD
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ME3183 administered orally for moderate to severe plaque psoriasis in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages 18 to 75 years
* Participant with stable moderate to severe chronic plaque psoriasis of at least 24 weeks duration.

Exclusion Criteria:

* Other than psoriasis, history of any clinically significant (as determined by the Investigator) or other major uncontrolled disease.
* Active or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at Screening.
* Hepatitis B surface antigen positive at Screening.
* History of HIV or Positive for the HIV antibodies at Screening.
* History of allergy to any component of the study treatment.
* Active tuberculosis (TB) or a history of incompletely treated TB.
* Active infection (bacteria, viral, fungal, etc.) requiring treatment with systemic antibiotics within 4 weeks of Screening.
* Malignancy or history of malignancy except for treated [ie, cured] basal cell or squamous cell in situ skin carcinomas and treated [ie, cured] cervical intraepithelial neoplasia or carcinoma in situ of the cervix with no evidence of recurrence.
* Pregnant or breast feeding
* Received ustekinumab, secukinumab, brodalumab, ixekizumab, guselkumab, risankizumab, tildrakizumab, or briakinumab within 24 weeks of first administration of study treatment.
* Received TNF-α inhibitor(s)/blocker(s) within 8 weeks of first administration of study treatment.
* Received rituximab within 24 weeks of first administration of study treatment.
* Received phototherapy or any systemic medications/treatments within 4 weeks of the first administration of study treatment.

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (14):
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - University of Southern California, Los Angeles, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - International Dermatology Research, INC, Miami, Florida
  - Qualmedica Research, LLC, Evansville, Indiana
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - Shondra L. Smith, MD Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Skin Search of Rochester, Inc., Rochester, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Studies in Dermatology, LLC, Cypress, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Center for Clinical Studies LTD, LLP, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (13):
  - Laser Rejuvenation Clinics Edmonton D.T. Inc, Edmonton, Alberta
  - SKiN Health, Cobourg, Ontario
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - Dermatrials Research Inc., Hamilton, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Dr. David Gratton Dermatologue Inc., Montreal, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2022 and concluded in May 2023.
Groups:
- ME3183 Dose 1, BID: Participants received ME3183 Dose 1 as a capsule along with matching placebo, twice daily for 16 weeks.
- ME3183 Dose 2, QD: Participants received ME3183 Dose 2 as a capsule along with matching placebo, once daily for 16 weeks.
- ME3183 Dose 3, BID: Participants received ME3183 Dose 3 as a capsule along with matching placebo, twice daily for 16 weeks.
- ME3183 Dose 4, QD: Participants received ME3183 Dose 4 as a capsule along with matching placebo, once daily for 16 weeks.
- Placebo: Participants received matching placebo of ME3183 as a capsule, twice daily for 16 weeks.
Period: Overall Study
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Started | 26 | 26 | 26 | 27 | 27
Completed | 17 | 14 | 18 | 15 | 16
Not Completed | 9 | 12 | 8 | 12 | 11
Not completed — Unacceptable toxicity or AE | 2 | 2 | 4 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 2 | 1
Not completed — Lost to Follow-up | 4 | 7 | 1 | 3 | 5
Not completed — Patient fails to adhere to the major protocol requirements | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who had signed Informed consent forms (ICFs) and had received a randomization number within the interactive web response system (IWRS) were included in the randomized set.
Groups:
- Total: Total of all reporting groups
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 26 | 27 | 27 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.42) | 46.2 (15.19) | 47.1 (14.60) | 45.7 (13.38) | 45.5 (16.54) | 46.3 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 7 | 12 | 48
  Male | 16 | 17 | 16 | 20 | 15 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 0 | 2 | 7 | 27
  Not Hispanic or Latino | 15 | 19 | 26 | 25 | 20 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 3 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 0 | 3
  White | 20 | 23 | 20 | 23 | 25 | 111
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 75% Reduction From Baseline in Psoriasis Area Severity Index (PASI) Score (PASI-75) at Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. The scores for each anatomic region are combined to yield the final PASI score.
  The final PASI score ranges from 0 to 72, with higher scores reflecting greater disease severity. Missing PASI at Week 16 are imputed as non-responders via NRI.
Time Frame: Week 16
Population: All participants who had been randomized, received at least 1 dose of the study drug and had at least 1 evaluable postbaseline time point were included in the Full analysis set (FAS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of participants | 58.3 [36.6 to 77.9] | 32.0 [14.9 to 53.5] | 61.5 [40.6 to 79.8] | 52.0 [31.3 to 72.2] | 14.8 [4.2 to 33.7]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Over the 16-week Treatment Period and the 4-week Follow-up Period
Description: An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening, worsens during the study, regardless of the suspected cause of the event. A Treatment-Emergent Adverse Event (TEAE) is an AE that occurred during the study after the first dose of study drug or that was present prior to dosing and exacerbates after the first dose of study drug.
Time Frame: Over the 16-week Treatment Period and the 4-week Follow-up Period (up to Week 20)
Population: All randomized participants who received at least 1 dose of study drug were included in the Safety Analysis Set (SAS). Analyses in the SAS were based on the study treatment received by each participant.
Measure: Count of Participants; unit: Participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 27
Participants | 16 | 17 | 23 | 24 | 16

3. Secondary Outcome: Number of Participants With Serious TEAEs Over the 16-week Treatment Period and the 4-week Follow-up Period
Description: An SAE is any untoward medical occurrence, in the view of either the investigator or Sponsor, that:
  * results in death,
  * is life-threatening,
  * results in inpatient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity, and/or
  * is a congenital anomaly/birth defect. Other important medical events that may not be immediately life-threatening or result in death or hospitalization, based upon appropriate medical judgement, are considered SAEs if they are thought to jeopardize the subject and/or require medical or surgical intervention to prevent one of the outcomes defining an SAE.
Time Frame: Over the 16-week Treatment Period and the 4-week Follow-up Period (up to Week 20)
Population: All randomized participants who received at least 1 dose of study drug were included in the SAS. Analyses in the SAS were based on the study treatment received by each participant.
Measure: Count of Participants; unit: Participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 27
Participants | 0 | 1 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With TEAEs by Severity Over the 16-week Treatment Period and the 4-week Follow-up Period
Description: An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening, worsens during the study, regardless of the suspected cause of the event. AEs were classified by severity as follows:
  MILD: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
  MODERATE: An event that is sufficiently discomforting to interfere with normal everyday activities.
  SEVERE: An event that prevents normal everyday activities.
Time Frame: Over the 16-week Treatment Period and the 4-week Follow-up Period (up to Week 20)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 27
Participants
  Mild | 7 | 11 | 8 | 15 | 11
  Moderate | 9 | 5 | 14 | 9 | 5
  Severe | 0 | 1 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: Physical Examination included height and body mass index. Any change in Physical examination abnormalities that were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: Over the 16-week Treatment Period and the 4-week Follow-up Period (up to Week 20)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 27
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs parameters included blood pressure, heart rate, respiratory rate, body temperature, and body weight. Any change in vital sign abnormalities that were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: Over the 16-week Treatment Period and the 4-week Follow-up Period (up to Week 20)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 27
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Tests
Description: Clinical laboratory testing included electrocardiogram (ECG), hematology, coagulation, blood chemistry, and urinalysis. Any change in clinical laboratory abnormalities that were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: Over the 16-week Treatment Period and the 4-week Follow-up Period (up to Week 20)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 27
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in PASI Score at All Visits From Week 1 to Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). Total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by degree of involvement for each anatomic region and then multiplied by constant. Scores for each anatomic region are combined to yield final PASI score (0 to 72). Higher scores= greater disease severity. Negative change from baseline indicates an improvement of disease symptoms. Percent reduction= (PASI score at Baseline - score at a follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: All participants who had been randomized, received at least 1 dose of the study drug and had at least 1 evaluable postbaseline time point were included in the FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Here, Number analyzed signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 23 | 24 | 23 | 25 | 27
percent change
  At Week 1: number analyzed (Participants) | 22 | 23 | 23 | 22 | 27
  At Week 1 | -22.87 (22.870) | -15.39 (21.708) | -24.47 (20.202) | -26.93 (26.966) | -12.01 (23.583)
  At Week 2: number analyzed (Participants) | 21 | 24 | 22 | 25 | 25
  At Week 2 | -42.41 (27.717) | -26.26 (24.172) | -41.91 (29.573) | -42.59 (24.412) | -18.44 (19.503)
  At Week 4: number analyzed (Participants) | 23 | 24 | 23 | 23 | 25
  At Week 4 | -47.82 (28.580) | -40.06 (30.657) | -56.77 (34.835) | -54.44 (26.596) | -21.55 (27.031)
  At Week 8: number analyzed (Participants) | 20 | 21 | 19 | 21 | 21
  At Week 8 | -66.38 (25.175) | -55.75 (28.436) | -83.31 (18.738) | -72.19 (22.642) | -24.17 (29.730)
  At Week 12: number analyzed (Participants) | 19 | 20 | 17 | 19 | 19
  At Week 12 | -72.31 (24.622) | -61.92 (29.350) | -87.22 (14.863) | -79.60 (18.063) | -36.18 (40.257)
  At Week 16: number analyzed (Participants) | 20 | 17 | 18 | 15 | 17
  At Week 16 | -74.77 (26.079) | -71.38 (25.923) | -90.77 (14.941) | -86.96 (12.414) | -40.26 (40.299)

9. Secondary Outcome: Percentage of Participants Achieving >=50% Reduction From Baseline in the PASI Score (PASI-50) at All Visits From Week 1 to Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by degree of involvement for each anatomic region and then multiplied by a constant. The scores for each anatomic region are combined to yield the final PASI score.
  The final PASI score ranges from 0 to 72, with higher scores reflecting greater disease severity. Missing PASI at Week 16 are imputed as non-responders via NRI.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: All participants who had been randomized, received at least 1 dose of the study drug and had at least 1 evaluable postbaseline time point were included in the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of participants
  At Week 1 | 12.5 [2.7 to 32.4] | 8.0 [1.0 to 26.0] | 7.7 [0.9 to 25.1] | 20.0 [6.8 to 40.7] | 7.4 [0.9 to 24.3]
  At Week 2 | 29.2 [12.6 to 51.1] | 8.0 [1.0 to 26.0] | 34.6 [17.2 to 55.7] | 36.0 [18.0 to 57.5] | 3.7 [0.1 to 19.0]
  At Week 4 | 50.0 [29.1 to 70.9] | 32.0 [14.9 to 53.5] | 61.5 [40.6 to 79.8] | 56.0 [34.9 to 75.6] | 14.8 [4.2 to 33.7]
  At Week 8 | 58.3 [36.6 to 77.9] | 52.0 [31.3 to 72.2] | 69.2 [48.2 to 85.7] | 64.0 [42.5 to 82.0] | 22.2 [8.6 to 42.3]
  At Week 12 | 70.8 [48.9 to 87.4] | 56.0 [34.9 to 75.6] | 61.5 [40.6 to 79.8] | 64.0 [42.5 to 82.0] | 33.3 [16.5 to 54.0]
  At Week 16 | 75.0 [53.3 to 90.2] | 52.0 [31.3 to 72.2] | 65.4 [44.3 to 82.8] | 60.0 [38.7 to 78.9] | 29.6 [13.8 to 50.2]

10. Secondary Outcome: Percentage of Participants Achieving >=75% Reduction From Baseline in the PASI Score (PASI-75) at All Visits From Week 1 to Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by degree of involvement for each anatomic region and then multiplied by a constant. The scores for each anatomic region are combined to yield the final PASI score.
  The final PASI score ranges from 0 to 72, with higher scores reflecting greater disease severity. Missing PASI at Week 16 are imputed as non-responders via NRI.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of participants
  At Week 1 | 4.2 [0.1 to 21.1] | 0 [0.0 to 13.7] | 0 [0.0 to 13.2] | 4.0 [0.1 to 20.4] | 0 [0.0 to 12.8]
  At Week 2 | 12.5 [2.7 to 32.4] | 8.0 [1.0 to 26.0] | 3.8 [0.1 to 19.6] | 8.0 [1.0 to 26.0] | 0 [0.0 to 12.8]
  At Week 4 | 20.8 [7.1 to 42.2] | 20.0 [6.8 to 40.7] | 34.6 [17.2 to 55.7] | 20.0 [6.8 to 40.7] | 3.7 [0.1 to 19.0]
  At Week 8 | 41.7 [22.1 to 63.4] | 20.0 [6.8 to 40.7] | 53.8 [33.4 to 73.4] | 52.0 [31.3 to 72.2] | 3.7 [0.1 to 19.0]
  At Week 12 | 45.8 [25.6 to 67.2] | 24.0 [9.4 to 45.1] | 57.7 [36.9 to 76.6] | 52.0 [31.3 to 72.2] | 14.8 [4.2 to 33.7]
  At Week 16 | 58.3 [36.6 to 77.9] | 32.0 [14.9 to 53.5] | 61.5 [40.6 to 79.8] | 52.0 [31.3 to 72.2] | 14.8 [4.2 to 33.7]

11. Secondary Outcome: Percentage of Participants Achieving >=90% Reduction From Baseline in the PASI Score (PASI-90) at All Visits From Week 1 to Week 16
Description: as for outcome 10
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of participants
  At Week 1 | 0 [0.0 to 14.2] | 0 [0.0 to 13.7] | 0 [0.0 to 13.2] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 2 | 0 [0.0 to 14.2] | 4.0 [0.1 to 20.4] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 4 | 4.2 [0.1 to 21.1] | 12.0 [2.5 to 31.2] | 7.7 [0.9 to 25.1] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 8 | 12.5 [2.7 to 32.4] | 16.0 [4.5 to 36.1] | 34.6 [17.2 to 55.7] | 16.0 [4.5 to 36.1] | 0 [0.0 to 12.8]
  At Week 12 | 20.8 [7.1 to 42.2] | 24.0 [9.4 to 45.1] | 34.6 [17.2 to 55.7] | 24.0 [9.4 to 45.1] | 3.7 [0.1 to 19.0]
  At Week 16 | 25.0 [9.8 to 46.7] | 20.0 [6.8 to 40.7] | 53.8 [33.4 to 73.4] | 28.0 [12.1 to 49.4] | 7.4 [0.9 to 24.3]

12. Secondary Outcome: Percentage of Participants Achieving 100% Reduction From Baseline in the PASI Score (PASI-100) at All Visits From Week 1 to Week 16
Description: as for outcome 10
Time Frame: Baseline, 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of participants
  At Week 1 | 0 [0.0 to 14.2] | 0 [0.0 to 13.7] | 0 [0.0 to 13.2] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 2 | 0 [0.0 to 14.2] | 4.0 [0.1 to 20.4] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 4 | 0 [0.0 to 14.2] | 8.0 [1.0 to 26.0] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 8 | 4.2 [0.1 to 21.1] | 8.0 [1.0 to 26.0] | 19.2 [6.6 to 39.4] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 12 | 4.2 [0.1 to 21.1] | 12.0 [2.5 to 31.2] | 19.2 [6.6 to 39.4] | 12.0 [2.5 to 31.2] | 0 [0.0 to 12.8]
  At Week 16 | 4.2 [0.1 to 21.1] | 20.0 [6.8 to 40.7] | 26.9 [11.6 to 47.8] | 16.0 [4.5 to 36.1] | 0 [0.0 to 12.8]

13. Secondary Outcome: Time to PASI-50
Description: Time to the first response of PASI-50 was defined as the number of days from the first dose of the study drug to the first response.
Time Frame: Baseline to Week 16
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
days | 33.5 [16.0 to 57.0] | 57.0 [29.0 to 86.0] | 28.0 [16.0 to 29.0] | 29.0 [15.0 to 43.0] | 113.0 [55.0 to NA] — Upper limit of 95% CI was not calculated due to less number of events.

14. Secondary Outcome: Time to PASI-75
Description: Time to the first response of PASI-75 was defined as the number of days from the first dose of the study drug to the first response.
Time Frame: Baseline to Week 16
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
days | 58.0 [55.0 to 111.0] | NA [57.0 to NA] — Median and Upper limit of 95% CI were not calculated due to less number of events. | 56.0 [29.0 to 61.0] | 57.0 [49.0 to 81.0] | NA [112.0 to NA] — Median and Upper limit of 95% CI were not calculated due to less number of events.

15. Secondary Outcome: Percentage of Participants Achieving a Static Physicians Global Assessment (sPGA) Score of "0" ("Clear") or "1" ("Almost Clear") Combined With 2-point Reduction on the 5-point sPGA Scale at All Visits From Week 1 to Week 16
Description: The Percentage of participants who achieved the static Physician's Global Assessment (sPGA) score of 'clear' or 'almost clear' (sPGA score 0 or 1) combined with 2-point reduction on the 5-point sPGA scale were reported. The investigator rated the severity of participant's psoriasis on the 5-point scale ranging from 0 (clear) to 4 (severe).
  0 = Clear: No signs of psoriasis. Post-inflammatory hyperpigmentation may be present.
  1. = Almost clear: Normal to pink coloration of lesions; no thickening; no to minimal focal scaling.
  2. = Mild: Pink to light red coloration; just detectable to mild thickening; predominantly fine scaling.
  3= Moderate: Dull bright red, clearly distinguishable erythema; clearly distinguishable to moderate thickening; moderate scaling.
  4 = Severe: Bright to deep dark red coloration; severe thickening with hard edges; severe/coarse scaling covering almost all or all lesions.
  Missing values are imputed as non-responders via NRI.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of participants
  At Week 1 | 0 [0.0 to 14.2] | 0 [0.0 to 13.7] | 0 [0.0 to 13.2] | 0 [0.0 to 13.7] | 0 [0.0 to 12.8]
  At Week 2 | 8.3 [1.0 to 27.0] | 8.0 [1.0 to 26.0] | 3.8 [0.1 to 19.6] | 4.0 [0.1 to 20.4] | 0 [0.0 to 12.8]
  At Week 4 | 4.2 [0.1 to 21.1] | 12.0 [2.5 to 31.2] | 19.2 [6.6 to 39.4] | 12.0 [2.5 to 31.2] | 0 [0.0 to 12.8]
  At Week 8 | 20.8 [7.1 to 42.2] | 12.0 [2.5 to 31.2] | 38.5 [20.2 to 59.4] | 36.0 [18.0 to 57.5] | 0 [0.0 to 12.8]
  At Week 12 | 29.2 [12.6 to 51.1] | 28.0 [12.1 to 49.4] | 42.3 [23.4 to 63.1] | 32.0 [14.9 to 53.5] | 7.4 [0.9 to 24.3]
  At Week 16 | 33.3 [15.6 to 55.3] | 32.0 [14.9 to 53.5] | 50.0 [29.9 to 70.1] | 28.0 [12.1 to 49.4] | 11.1 [2.4 to 29.2]

16. Secondary Outcome: Change From Baseline in Affected Body Surface Area (BSA) at All Visits From Week 1 to Week 16
Description: BSA is a measurement of the affected skin area. The overall BSA affected by psoriasis plaques is estimated based on the palm area of the participant hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total BSA. Negative change from baseline indicates improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of body surface area
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
percentage of body surface area
  At Week 1 | -1.6 [-3.9 to 0.7] | -2.1 [-4.3 to 0.1] | -3.6 [-5.8 to -1.4] | -3.5 [-5.7 to -1.2] | -0.8 [-2.9 to 1.3]
  At Week 2 | -5.6 [-8.2 to -2.9] | -3.6 [-6.2 to -1.1] | -6.7 [-9.3 to -4.1] | -4.7 [-7.2 to -2.1] | -1.9 [-4.4 to 0.5]
  At Week 4 | -6.9 [-9.8 to -4.0] | -6.2 [-9.1 to -3.4] | -9.5 [-12.4 to -6.7] | -7.3 [-10.1 to -4.4] | -2.6 [-5.4 to 0.2]
  At Week 8 | -12.2 [-15.6 to -8.7] | -9.0 [-12.4 to -5.7] | -15.3 [-18.7 to -11.8] | -11.8 [-15.1 to -8.4] | -3.6 [-6.8 to -0.4]
  At Week 12 | -15.1 [-18.8 to -11.4] | -11.9 [-15.5 to -8.3] | -16.7 [-20.5 to -12.9] | -12.9 [-16.6 to -9.3] | -4.4 [-8.0 to -0.9]
  At Week 16 | -16.4 [-20.4 to -12.4] | -12.1 [-16.1 to -8.0] | -17.3 [-21.4 to -13.1] | -14.4 [-18.6 to -10.3] | -7.6 [-11.6 to -3.6]

17. Secondary Outcome: Change From Baseline in the Itch Numerical Rating Scale (NRS) at All Visits From Week 1 to Week 16
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." The overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours. Negative change from baseline indicates improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
score on a scale
  At Week 1 | -1.7 [-2.6 to -0.8] | -1.5 [-2.3 to -0.6] | -2.7 [-3.5 to -1.8] | -2.3 [-3.2 to -1.5] | -1.2 [-2.0 to -0.4]
  At Week 2 | -3.3 [-4.3 to -2.3] | -2.1 [-3.0 to -1.2] | -3.0 [-3.9 to -2.1] | -3.3 [-4.2 to -2.4] | -0.7 [-1.6 to 0.2]
  At Week 4 | -2.9 [-4.0 to -1.8] | -2.7 [-3.8 to -1.7] | -3.9 [-4.9 to -2.8] | -3.7 [-4.8 to -2.7] | -0.5 [-1.5 to 0.5]
  At Week 8 | -4.0 [-5.1 to -2.9] | -3.6 [-4.6 to -2.6] | -4.6 [-5.7 to -3.6] | -4.4 [-5.4 to -3.4] | -1.0 [-2.0 to 0.0]
  At Week 12 | -4.4 [-5.5 to -3.3] | -3.9 [-4.9 to -2.8] | -4.9 [-6.0 to -3.8] | -4.0 [-5.1 to -3.0] | -1.4 [-2.5 to -0.4]
  At Week 16 | -4.8 [-5.9 to -3.7] | -3.9 [-5.0 to -2.8] | -5.0 [-6.1 to -3.9] | -4.5 [-5.6 to -3.3] | -1.4 [-2.5 to -0.3]

18. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Score at All Visits From Week 1 to Week 16
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on a participant's quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI a total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on the quality of life of participants. Negative change from baseline indicates improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 24 | 25 | 26 | 25 | 27
score on a scale
  At Week 1 | -2.2 [-4.2 to -0.3] | -2.4 [-4.2 to -0.5] | -5.0 [-6.8 to -3.2] | -3.3 [-5.1 to -1.4] | -4.1 [-5.8 to -2.4]
  At Week 2 | -5.1 [-7.0 to -3.1] | -5.6 [-7.5 to -3.8] | -6.2 [-8.0 to -4.3] | -5.5 [-7.3 to -3.6] | -3.4 [-5.2 to -1.6]
  At Week 4 | -5.2 [-7.4 to -3.0] | -6.0 [-8.2 to -3.9] | -8.1 [-10.2 to -6.0] | -6.4 [-8.5 to -4.2] | -3.4 [-5.5 to -1.4]
  At Week 8 | -6.9 [-9.1 to -4.7] | -6.4 [-8.5 to -4.2] | -8.8 [-11.0 to -6.6] | -8.0 [-10.2 to -5.9] | -4.0 [-6.1 to -2.0]
  At Week 12 | -7.8 [-10.1 to -5.6] | -6.2 [-8.4 to -4.1] | -9.5 [-11.7 to -7.2] | -8.9 [-11.1 to -6.7] | -3.6 [-5.7 to -1.5]
  At Week 16 | -8.3 [-10.3 to -6.3] | -6.9 [-8.9 to -5.0] | -9.6 [-11.5 to -7.6] | -9.5 [-11.5 to -7.5] | -3.7 [-5.7 to -1.8]

19. Secondary Outcome: Percentage of Participants With at Least a 5-point Reduction From Baseline in the DLQI Score at All Visits From Week 1 to Week 16
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on a participant's quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI a total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on the quality of life of participants.
Time Frame: Baseline, Week 1, 2, 4, 8, 12 and 16
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
Number analyzed (Participants) | 22 | 24 | 23 | 25 | 27
percentage of participants
  At Week 1: number analyzed (Participants) | 21 | 23 | 23 | 22 | 27
  At Week 1 | 22.7 [7.8 to 45.4] | 26.1 [10.2 to 48.4] | 65.2 [42.7 to 83.6] | 36.4 [17.2 to 59.3] | 44.4 [25.5 to 64.7]
  At Week 2: number analyzed (Participants) | 20 | 24 | 22 | 25 | 25
  At Week 2 | 52.4 [29.8 to 74.3] | 41.7 [22.1 to 63.4] | 63.6 [40.7 to 82.8] | 56.0 [34.9 to 75.6] | 36.0 [18.0 to 57.5]
  At Week 4: number analyzed (Participants) | 22 | 24 | 23 | 23 | 25
  At Week 4 | 47.8 [26.8 to 69.4] | 41.7 [22.1 to 63.4] | 60.9 [38.5 to 80.3] | 56.5 [34.5 to 76.8] | 40.0 [21.1 to 61.3]
  At Week 8: number analyzed (Participants) | 19 | 21 | 19 | 21 | 22
  At Week 8 | 60.0 [36.1 to 80.9] | 47.6 [25.7 to 70.2] | 68.4 [43.4 to 87.4] | 81.0 [58.1 to 94.6] | 50.0 [28.2 to 71.8]
  At Week 12: number analyzed (Participants) | 19 | 20 | 17 | 19 | 19
  At Week 12 | 55.0 [31.5 to 76.9] | 50.0 [27.2 to 72.8] | 82.4 [56.6 to 96.2] | 78.9 [54.4 to 93.9] | 42.1 [20.3 to 66.5]
  At Week 16: number analyzed (Participants) | 19 | 17 | 18 | 15 | 17
  At Week 16 | 60.0 [36.1 to 80.9] | 58.8 [32.9 to 81.6] | 77.8 [52.4 to 93.6] | 93.3 [68.1 to 99.8] | 35.3 [14.2 to 61.7]

20. Secondary Outcome: Trough Serum Concentration (Ctrough) of ME3183
Description: Ctrough of study drug was determined from the plasma samples using a validated analytical method.
Time Frame: Pre-dose at Week 1, 4, 8 and 16
Population: The PK analysis set consisted of all participants who were correctly administered at least 1 ME3183 dose and where ME3183 concentration data is available without any protocol deviation interfering with these results. Analyses in PK analysis set was based on the study treatment actually received by each participant. Here, number of participants analyzed= participants who were evaluable for this outcome measure. Number analyzed= participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per liter (ng/L)
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD
Number analyzed (Participants) | 19 | 18 | 18 | 18
nanograms per liter (ng/L)
  At Week 1: number analyzed (Participants) | 16 | 18 | 18 | 18
  At Week 1 | 13998.33 (88.57) | 11491.05 (82.48) | 28559.81 (55.62) | 21229.09 (78.54)
  At Week 4: number analyzed (Participants) | 19 | 16 | 17 | 13
  At Week 4 | 17973.10 (53.45) | 16522.41 (63.92) | 24920.33 (139.68) | 25396.74 (102.98)
  At Week 8: number analyzed (Participants) | 16 | 15 | 17 | 10
  At Week 8 | 14606.67 (49.37) | 13046.98 (73.86) | 27970.28 (82.55) | 16320.92 (162.08)
  At Week 16: number analyzed (Participants) | 10 | 10 | 14 | 9
  At Week 16 | 10616.79 (78.77) | 11444.51 (227.49) | 23327.81 (72.11) | 9081.21 (454.97)

ADVERSE EVENTS:
Time Frame: From Baseline up to the end of the Follow-up Period (up to Week 20)
Description: A TEAE is an AE that occurs during the study after the first dose of the study drug or that is present before dosing and exacerbates after the first dose of the study drug.
Arm/Group | ME3183 Dose 1, BID | ME3183 Dose 2, QD | ME3183 Dose 3, BID | ME3183 Dose 4, QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/26 | 0/26 | 0/26 | 1/27
Other Adverse Events (participants affected / at risk) | 10/25 | 14/26 | 20/26 | 21/26 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ME3183 Dose 1, BID (N=25) | ME3183 Dose 2, QD (N=26) | ME3183 Dose 3, BID (N=26) | ME3183 Dose 4, QD (N=26) | Placebo (N=27)
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ME3183 Dose 1, BID (N=25) | ME3183 Dose 2, QD (N=26) | ME3183 Dose 3, BID (N=26) | ME3183 Dose 4, QD (N=26) | Placebo (N=27)
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 8 | 10 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 8 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 2 | 2
COVID-19 (Infections and infestations) | 0 | 1 | 3 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 2 | 11 | 7 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 2 | 0
Lipase increased (Investigations) | 1 | 0 | 4 | 3 | 1
Blood pressure increased (Investigations) | 0 | 0 | 3 | 4 | 0
Weight decreased (Investigations) | 0 | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT05268016/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT05268016/SAP_001.pdf